CLINICAL TRIAL: NCT02440880
Title: Dexamethasone With TAP Block Increasing the Duration of the Peripheral Nerve Block in Caesarian Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hassan Mohamed Ali, lecturer in anesthesia department Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Qasr Elainy
Record Dates: First submitted 2015-04-24; First posted 2015-05-12 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Dexamethasone; Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- CONTROL (Placebo Comparator): TAP block without Dexamethasone neither intravenous nor in combination with the block
  Interventions: Other: control
- Group 2 (TD8IS) (Experimental): Dexamethasone in combination with TAP block in dose of 8 mg
  Interventions: Drug: Dexamethasone in combination with TAP block in dose of 8 mg
- Group 3(TD4IS) (Experimental): Dexamethasone in addition to TAP block in dose of 4 mg
  Interventions: Drug: Dexamethasone in addition to TAP block in dose of 4 mg
- Group 4 (TSID8): (Experimental): Dexamethasone intravenous in addition to TAP block in dose of 8 mg
  Interventions: Drug: Dexamethasone intravenous in addition to TAP block in dose of 8 mg
- Group5(TSID4) (Experimental): Dexamethasone intravenous 4mg+ TAP block
  Interventions: Drug: Dexamethasone intravenous 4mg+ TAP block

INTERVENTIONS:
Drug: Dexamethasone in addition to TAP block in dose of 4 mg — Dexamethasone in addition to TAP block in dose of 4 mg
  Arms: Group 3(TD4IS)
Drug: Dexamethasone in combination with TAP block in dose of 8 mg — Dexamethasone in combination with TAP block in dose of 8 mg
  Arms: Group 2 (TD8IS)
Drug: Dexamethasone intravenous 4mg+ TAP block — Dexamethasone intravenous in addition to TAP block in dose of 4 mg
  Other Names: Dexamethasone intravenous 4mg + TAP block
  Arms: Group5(TSID4)
Drug: Dexamethasone intravenous in addition to TAP block in dose of 8 mg — Dexamethasone intravenous + TAP block in dose of 8 mg
  Other Names: Dexamethasone intravenous 8mg+ TAP block
  Arms: Group 4 (TSID8):
Other: control — TAP block without Dexamethasone neither intravenous nor in combination with the block
  Other Names: control group
  Arms: CONTROL

SUMMARY:
Nowadays Cesarean sections became the most popular surgery worldwide with the consumption of the hospital resources and the continuous need to decrease the costs, work load and medical stuff engagement. One of the most common problem is the need to control pain post operatively, this issue increase the work load over the pain management team and increase lead to patient in satisfaction.

This study will test the usage of dexamethasone with different doses (4 and 8 mg) either locally or intravenously (I.V.) with the local anesthetics in TAP (transversus abdominis plane) block to prolong the duration of the block and decrease the need of post-operative analgesics.

DETAILED DESCRIPTION:
Nowadays Cesarean sections became the most popular surgery worldwide with the consumption of the hospital resources and the continuous need to decrease the costs, work load and medical stuff engagement. One of the most common problem is the need to control pain post operatively, this issue increase the work load over the pain management team and increase lead to patient in satisfaction.(1,2,3) The presence of the adjuvant which can be added to the conventional anesthetic medications can prolong the duration of action and decrease the need for frequent post-operative analgesics.(4,5) The idea of adding a catheter or placing an epidural catheter still have a quite limitation regarding the patients compliance, delayed ambulation and high costs, these limitations redirect the anesthetist again to the use of adjuvant with a single shot block to prolong the duration of it and decrease the need of subsequent analgesics.(6) Dexamethasone proved to be an effective adjuvant in prolongation of the nerve blocks with the question regarding the proper route and dose (7,8,9,10).

This study will test the usage of dexamethasone with different doses (4 and 8 mg) either locally or intravenously (I.V.) with the local anesthetics in TAP (transversus abdominis plane) block to prolong the duration of the block and decrease the need of post-operative analgesics.

ELIGIBILITY:
Inclusion Criteria:

* Any patient ASA (american society of anesthesia) I or II,
* aged between 18 and 45 scheduled for elective cesarean section.

Exclusion Criteria:

* patient refusal,
* age below 18 or above 45 years,
* coagulopathy with INR (international normalized ratio) more than 1.5 or platelets below 100000,
* uncontrolled diabetes, uncontrolled hypertensive, addict patient,
* psychological instability, and
* allergy to the used drugs,
* failure of spinal,
* conversion to general of anesthesia,
* failure of application of TAP block.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-11 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
level of pain according to verbal analogue scale | THREE DAYS

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Ali, LECTURER, Principal Investigator — Anesthesia department, faculty of medicine ,Cairo university
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided